CLINICAL TRIAL: NCT00002599
Title: MYELOMA VII MEDICAL RESEARCH COUNCIL WORKING PARTY ON LEUKEMIA IN ADULTS: MYELOMATOSIS THERAPY TRIAL
Brief Title: Combination Chemotherapy and Interferon Alfa With or Without Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Myeloma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063834; MRC-LEUK-MYEL-VII; EU-94030
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Filgrastim; Interferon-alpha; sargramostim; Carmustine; Cyclophosphamide; Doxorubicin; Melphalan; Methylprednisolone; Prednisone; Vincristine

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Biological: sargramostim
Drug: carmustine
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: melphalan
Drug: methylprednisolone
Drug: prednisone
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bone marrow or peripheral stem cell transplantation with chemotherapy may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Interferon alfa may interfere with the growth of cancer cells. It is not yet known whether a more intensive chemotherapy regimen plus stem cell or bone marrow transplant is more effective than standard chemotherapy in treating patients with myeloma.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of combination chemotherapy plus interferon alfa with or without high dose melphalan or bone marrow or peripheral stem cell transplantation in treating patients with previously untreated myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival of patients under age 65 with myeloma treated with standard ABCM (doxorubicin, carmustine, cyclophosphamide, melphalan) vs. intensive C-VAMP (cyclophosphamide, vincristine, doxorubicin, methylprednisolone) followed by high-dose melphalan (with or without total-body irradiation) with bone marrow and peripheral blood stem cell support, both with IFN-A maintenance. II. Compare the toxicity profiles of the 2 treatment arms. III. Compare the 2 treatment arms with respect to quality of life and health economics issues. IV. Investigate cellular changes by means of linked morphology, phenotype, and cytogenetics studies before and after treatment and at relapse.

OUTLINE: Randomized study. The following acronyms are used: ABM Autologous Bone Marrow BCNU Carmustine, NSC-409962 CTX Cyclophosphamide, NSC-26271 DOX Doxorubicin, NSC-123127 G-CSF Granulocyte Colony Stimulating Factor (Amgen), NSC-614629 GM-CSF Granulocyte-Macrophage Colony Stimulating Factor (source not specified) IFN-A Interferon alpha (Hoffmann-La Roche), NSC-367982 L-PAM Melphalan, NSC-8806 MePRDL Methylprednisolone, NSC-19987 PBSC Peripheral Blood Stem Cells PRED Prednisone, NSC-10023 TBI Total-Body Irradiation VCR Vincristine, NSC-67574 ARM I. Induction: 4-Drug Combination Chemotherapy or, as indicated, 2-Drug Combination Chemotherapy. ABCM: DOX; BCNU; CTX; L-PAM; or, if pretreatment ANC and platelets are less than 1,300 and 75,000, CTX; PRED. Maintenance: Biological Response Modifier Therapy. IFN-A. ARM II. Induction: 4-Drug Combination Chemotherapy followed by Hematopoietic Stimulation. C-VAMP: DOX; VCR; MePRDL; CTX; followed by CTX; G-CSF or GM-CSF. Consolidation: 3-Drug Combination Chemoablation with or without Radioablation followed by Hematopoietic Rescue. CTX; L-PAM; MePRDL; with or without TBI using megavoltage equipment (linear accelerator preferred); followed by ABM and/or PBSC. Maintenance: Biological Response Modifier Therapy. IFN-A.

PROJECTED ACCRUAL: 750 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Definite myeloma requiring chemotherapy and fulfilling at least 2 of the following criteria: Neoplastic plasma cell infiltrate and/or microplasmacytomas on bone marrow aspiration and/or trephine Paraprotein in blood and/or urine Definite lytic bone lesions (not simply osteoporosis) No equivocal myeloma (such patients should be registered with the Clinical Trial Service Unit, Oxford)

PATIENT CHARACTERISTICS: Age: Under 65 Performance status: Not specified Hematopoietic: (following rehydration and treatment for infection, if necessary) ANC at least 1,000 Platelets at least 50,000 Hepatic: Not specified Renal: Renal insufficiency does not necessarily exclude (dose reduction may be applicable) Cardiovascular: No severe cardiac disease Past history of ischemic heart disease may exclude at the discretion of the investigator Pulmonary: No severe respiratory illness Other: Ability to tolerate at least 3 liters/day of fluid No life-threatening disease unrelated to myeloma Prior or concurrent psychiatric disorder may exclude at the discretion of the investigator No prior malignancy except: Nonmelanomatous skin tumors In situ carcinomas

PRIOR CONCURRENT THERAPY: No prior therapy other than minimal local radiotherapy for relief of bone pain

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 1994-09

CONTACTS AND LOCATIONS:
Overall Officials: J. A. Child, MD, Study Chair — Leeds General Infirmary
Locations (1):
- Leeds Teaching Hospital Trust, Leeds, England, United Kingdom